CLINICAL TRIAL: NCT03133117
Title: Deficits, Adaptation and Cerebral Functional Reorganization of Visual Retinotopic Treatments During Normal and Pathological Aging (Age-related Macular Degeneration and Glaucoma)
Acronym: VISIOPERICENT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC16.070
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Macular Degeneration; Glaucoma
MeSH Terms: conditions — Macular Degeneration; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebral Bases of Central and Peripheral Visual Integration (Experimental)
  Interventions: Radiation: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Radiation: Functional Magnetic Resonance Imaging (fMRI) — Functional Magnetic Resonance Imaging (fMRI)

SUMMARY:
The main objective of this research is to study the cognitive and cerebral mechanisms of the integration of central and peripheral visual information during normal and pathological aging (ophthalmological patients with AMD and glaucoma) through fMRI studies. To assess the effect of normal aging, research will be conducted on a group of young participants with normal vision and a group of elderly participants with normal vision. Each participant will be assessed once during an MRI (during which the brain activity and behavioral performance will be measured). In order to evaluate the effect of pathological aging, research will be conducted on AMD patients, glaucomatous patients, and age-matched controls (normal vision), evaluated only once during an MRI examination.

DETAILED DESCRIPTION:
Healthy / control participants with normal vision will be volunteers, selected after interview (inclusion assessment). Their recruitment will be carried out on the basis of advertisements displayed at Grenoble Alpes University. Patients will be volunteers, selected on the basis of their ophthalmological clinical record. Their recruitment will be done at the Ophthalmology Clinic of the University Hospital of Grenoble (through Professor Florent Aptel). For all the participants, a medical examination before MRI examination will be carried out in the MRU unit of the CHU of Grenoble in order to verify the eligibility criteria for contraindications to MRI and MRI scanning. The results of these examinations will be communicated to the subjects prior to the expression of their consent directly or through the doctor of their choice.

ELIGIBILITY:
Inclusion Criteria:

* Healthy / control participants: normal or normal corrected visual acuity
* Patients with AMD: Diagnosis of AMD by the Clinique d'ophtalmologie of the CHU de Grenoble
* Patients Glaucoma: Diagnosis of glaucoma by the Clinique d'ophtalmologie of the CHU de Grenoble
* Affiliation to a social security scheme,
* Informed consent signed,
* Medical examination before participation in the MRI examination

Exclusion Criteria:

* Major unprotected persons unable to express their consent,
* Major protected,
* Significant hearing impairment,
* Neuropsychiatric pathology past or present (except benign epilepsy),
* Taking narcotics and / or drugs for neurocognitive purposes,
* Existence of a general ailment (cardiac, respiratory, haematological, renal, hepatic, cancer),
* Other ophthalmic pathology that can affect visual function: cataract, retinal detachment
* Contra-indication to MRI:

  1. Any subject with a vascular stent implanted less than 6 weeks before the examination.
  2. Any subject carrying implanted biomedical material judged "unsafe" or "unsafe" in the list: http://www.mrisafety.com/TheList_search.asp.
  3. Any acquisition procedure that does not comply with the conditions required by the "conditional" use in a subject carrying implanted biomedical material considered "conditional" in the list: http://www.mrisafety.com/TheList_search. Asp.
  4. Any subject carrying an intra-ocular or intracranial ferromagnetic foreign body close to the nervous structures.
  5. Any subject with biomedical equipment such as a cardiac, neuronal or sensory pacemaker (cochlear implant) or a ventricular bypass valve without medical and paramedical support trained to perform MRI in these subjects.
  6. Non-Cooperative Subject
  7. Metallic or electronic equipment incompatible with MRI examination, dental apparatus, claustrophobia, pacemaker or neurologic, non-magnetic non-magnetic vascular clip, metallic luster, diabetes
* Pregnant women
* Woman of childbearing age refusing to take the pregnancy test
* Ongoing drug treatment that may affect brain activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Accuracy of visual tasks in relation to the intensity of cerebral activity measured in fMRI | One hour
  Measurement of cerebral activity during visual tasks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Ophtalmologique Universitaire de Grenoble, Grenoble, CHU Albert Michallon - CS 10217, France